CLINICAL TRIAL: NCT04078438
Title: Neurofeedback Treatment on Depressive Symptoms and Functional Recovery in Treatment-resistant Patients With Major Depressive Disorder: an Open-label Pilot Study
Brief Title: Neurofeedback In Treatment Resistant Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of researcher foreign training
Sponsor: Yeungnam University Hospital (Other)
Responsible Party: Principal Investigator, Eun-Jin Cheon, Principal Investigator, Yeungnam University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: YUH-14-0389-B4
Record Dates: First submitted 2019-08-22; First posted 2019-09-06 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Depression; Neurofeedback
Keywords: Treatment-resistant depression; Neurofeedback; Functional recovery
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant | interventions — Therapeutics; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- neurofeedback augmentation group (Experimental): The neurofeedback augmentation group was asked to participate in 12 weeks of combined therapy of medication and 12-24 sessions of neurofeedback training. The neurofeedback protocol was determined considering the patient's main symptoms. Patients in the neurofeedback augmentation group received sensorimotor rhythm (SMR) beta or beta training for 30 minutes, and then alpha/theta (A/T) training for 30 minutes in each session.
  Interventions: Device: neurofeedback augmentation; Drug: treatment as usual
- medication-only (treatment as usual, TAU) group (Active Comparator): To reduce the impact of confounding factors, the medication-only (treatment as usual, TAU) group visited at the same schedule as neurofeedback augmentation group and received psychotherapy placebo sessions instead of neurofeedback training sessions. These sessions included psychological assessment and supportive psychotherapy. The medication-only (treatment as usual, TAU) group maintained the same medication use as that before the study.
  Interventions: Drug: treatment as usual; Other: psychotherapy placebo sessions
- healthy controls (No Intervention): The healthy controls provided blood samples using the same procedure at baseline only.

INTERVENTIONS:
Device: neurofeedback augmentation — Neurofeedback training was performed using a Neurocybernetics EEG Biofeedback system (Neurocybernetics Inc., Encino, CA, USA). The neurofeedback protocol was determined by the neurofeedback team, which included 3 psychiatrists, in consideration of the patient's main symptoms.
  The neurofeedback augmentation group was asked to participate in 12 weeks of combined therapy of medication and 12-24 sessions of neurofeedback training. Patients in the neurofeedback augmentation group received sensorimotor rhythm (SMR) beta or beta training for 30 minutes, and then alpha/theta (A/T) training for 30 minutes in each session.
  To reduce the impact of confounding factors, the medication-only (treatment as usual, TAU) group visited at the same schedule as neurofeedback augmentation group and received psychotherapy placebo sessions. The medication-only (treatment as usual, TAU) group maintained the same medication use as that before the study.
  Arms: neurofeedback augmentation group
Drug: treatment as usual — The neurofeedback augmentation group and the medication-only group maintained the same medication use as that before the study.
  Other Names: medication
  Arms: medication-only (treatment as usual, TAU) group; neurofeedback augmentation group
Other: psychotherapy placebo sessions — To reduce the impact of confounding factors, the medication-only (treatment as usual, TAU) group visited at the same schedule as neurofeedback augmentation group and received psychotherapy placebo sessions instead of neurofeedback training sessions. These sessions included psychological assessment and supportive psychotherapy.
  Arms: medication-only (treatment as usual, TAU) group

SUMMARY:
The investigators evaluate the effects of neurofeedback as an augmentation treatment on depressive symptoms and functional recovery in patients with treatment-resistant depression (TRD).

TRD patients are assigned to the neurofeedback augmentation group and the medication-only (treatment as usual, TAU) group. The neurofeedback augmentation group underwent combined therapy comprising medication and 12-24 sessions of neurofeedback training for 12 weeks. To assess the serum levels of brain-derived neurotrophic factor (BDNF) in both groups, a pre- and post-treatment blood samples are obtained. Patients are evaluated using the Hamilton Depression Rating Scale (HAM-D), Beck Depression Inventory (BDI), Clinical Global Impression-Severity (CGI-S), 5-level version of European Quality of Life Questionnaire 5-Dimensional Classification (EQ-5D-5L), and Sheehan Disability Scale (SDS) at baseline, and at the 1-, 4-, and 12-week.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a severely disabling disorder resulting in the deterioration of daily function and lowering quality of life. The lifetime prevalence of depression is 10-15%, and the annual prevalence of MDD in the United States is approximately 7%. The World Health Organization has reported that MDD is expected to be the top disease in terms of global burden by 2030. Fifty percent of patients with depressive disorder have a chronic disease course, and 20% of such patients have insufficient responses to treatment despite the use of antidepressant medication. In addition, although antidepressants have been shown to be effective, residual symptoms may continue by stopping the medication early due to inconvenient side effects of the medication. Sixty percent of patients with depressive disorder have poorer executive function. Patients with depressive disorder are continuously affected by deficits in social functioning, such as interpersonal relationships and job adaptation, even if some of their symptoms are improved by medication. Therefore, various additional treatments other than antidepressant treatment have been tried to improve residual depressive symptoms and the remission rate.

Brain waves have been used to measure brain activity and previous studies have reported that different brain waves reflect different brain states, including moods. Neurofeedback is a type of electroencephalography (EEG) training that allows individuals to change the levels of particular types of brain waves displayed on a computer by operational conditioning. EEG studies showed that the neurofeedback is capable of generating long term changes in the spectral EEG topography, while neuroimaging studies represented the neuroplastic effects from neurofeedback treatment. Neurofeedback is an alternative approach that aims to help individuals alter brain activation without introducing electrical or magnetic activity, or pharmacological compounds into the brain, hence preventing the brain from becoming dependent on outside influences for better functioning. It is noninvasive method and there's no report of even minor side effects.

Neurofeedback may be considered a new augmentation treatment for patients with treatment-resistant depression (TRD), even after the use of antidepressants. Some studies have reported improvements in both depressive symptoms and executive function following neurofeedback treatment. A recent article insisted that neurofeedback treatment for depression as having "revealed promising effects in recent clinical trials". However, most such studies have been case reports or uncontrolled studies, and the mechanism underlying the treatment effects of neurofeedback are still unclear. In addition, there has been no study of neurofeedback on depressive symptoms and functional recovery in patients with TRD.

Brain-derived neurotrophic factor (BDNF) acts on certain neurons of the central nervous system and the peripheral nervous system. It helps support the survival of existing neurons and encourages the growth and differentiation of new neurons and synapses. Previous studies have suggested the presence of an etiological link between the development of depression and BDNF. However, no studies have examined the association between neurofeedback and changes in BDNF level.

The purpose of this pilot study was to evaluate the effects of neurofeedback as an augmentation treatment on depressive symptoms and functional recovery in patients with TRD. The investigators also aimed to identify the usefulness of BDNF as a biomarker for neurofeedback by examining changes in the BDNF level before vs. after treatment in the neurofeedback treatment and medication-only (treatment as usual, TAU) groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagosis with MDD according to the DSM-IV-TR criteria for MDD, and especially treatment-resistant MDD (Hamilton Rating Scale for Depression [HAM-D] score ⩾14) despite adequate antidepressant therapy)

Exclusion Criteria:

* Psychosis
* Bipolar disorder
* Brain injury
* Clinically diagnosed neurological disorder
* Convulsive disorder
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-02-08 (Actual)

PRIMARY OUTCOMES:
Changes in Hamilton Rating Scale for Depression [HAM-D] score at baselline and the 1-, 4-, and 12-week time points | at baseline, and at the 1-, 4-, and 12-week time points.
  The HAM-D is an observer rating scale and 1 of the most widely used measures of depressive disorder. This scale composed of 17 items, and it has been used to assess the therapeutic effect as well as the severity of depression. Total score is 52, where higher scores indicating more severe depression. Hamilton considered Total score of 8-13 mild range, 14-18 moderate, 18-22 severe, and 23 or higher very severe.

SECONDARY OUTCOMES:
Changes in Beck Depression Inventory- II (BDI-II) scores at baselline and the 1-, 4-, and 12-week time points | at baseline, and at the 1-, 4-, and 12-week time points.
  The BDI is self-report scale designed to evaluate the presence and severity of depressive symptoms. It is consisted of 21 items including cognitive, emotional, motivative, and physical symptoms of depression. Each question is scored from 0 to 3 points, and the total score ranges from 0 to 63, indicating the higher the total scores, the more severe the depression. It is considered total score of 0-9 minimal range, 10-15 mild, 16-23 moderate, and 24-63 severe.
Changes in Sheehan Disability Scale (SDS) score at baselline and the 1-, 4-, and 12-week time points | at baseline, and at the 1-, 4-, and 12-week time points.
  The SDS is a self-report scale designed by Sheehan to assess the severity of functional impairment. This scale consists of 3 items, and each item is divided into 11 levels from 0 to 10 points. It is considered 0 point: none, 1-3 points: mild, 4-6 points: moderate, and 7-10 points: severe. Total score ranges from 0 to 30 and means that the higher the total scores, the more severe the functional impairment.
Changes in Clinical Global Impression-Severity (CGI-S) at baselline and the 1-, 4-, and 12-week time points | at baseline, and at the 1-, 4-, and 12-week time points.
  The CGI-S is a single-item scale composed of 7 levels ranging from maximum score of 7 to normal state of 1. This scale is a measure by which the evaluator comprehensively assesses the severity of mental illness regardless of diagnosis.
Comparisons of serum brain-derived neurotrophic factor (BDNF) level between baseline and the 12-week time point among groups | at baseline, and 12-week time points.
  Brain-derived neurotrophic factor (BDNF) acts on certain neurons of the central nervous system and the peripheral nervous system. It helps support the survival of existing neurons and encourages the growth and differentiation of new neurons and synapses. Previous studies have suggested the presence of an etiological link between the development of depression and BDNF.
Type and number of adverse events | through study completion, an average of 12 weeks
  adverse events
Changes in valuation of 5 level version of European Quality of Life Questionnaire 5-Dimensional Classification (EQ-5D-5L) (converted tariff score) | at baseline, and at the 1-, 4-, and 12-week time points.
  The EQ-5D-5L was developed by the EuroQol Group, and is used to assess 5 dimensions: mobility, self care, usual activity, pain/discomfort, and anxiety/depression. Each dimension is consisted of 5 levels, so total 3125 health states can be evaluated. The valuation of EQ-5D-5L (converted tariff score) is an index score calculated by applying weight to each of the 5 EQ-5D-5L questionnaires to provide a comprehensive summary of health-related quality of life. The resulting set of tariff is widely used to calculate preferences for EQ-5D-5L health states. As EQ-5D-5L is translated according to the culture and situation of each country, EQ-5D-5L tariffs may differ at each country. The index score is valued from 0 to 1, and the higher scores indicate the higher quality of life for the patients. In this study, EQ-5D-5L tariffs (index values) were calculated according to the [The EQ-5D-5L valuation study in Korea.].
Changes in response and remission rate of Hamilton Rating Scale for Depression [HAM-D] score | at baseline, and at the 1-, 4-, and 12-week time points.
  Remission was defined as achieving a HAM-D score below 7, and response was defined as a 50% or greater reduction in HAM-D score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Jin Cheon, M.D., Ph.D, Study Director — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

REFERENCES:
- [Derived] Lee YJ, Lee GW, Seo WS, Koo BH, Kim HG, Cheon EJ. Neurofeedback Treatment on Depressive Symptoms and Functional Recovery in Treatment-Resistant Patients with Major Depressive Disorder: an Open-Label Pilot Study. J Korean Med Sci. 2019 Nov 4;34(42):e287. doi: 10.3346/jkms.2019.34.e287. PMID 31674161